CLINICAL TRIAL: NCT06164769
Title: A Prospective Study of Enucleation of Pancreatic Tumor by Blocking Abdominal Trunk and Superior Mesenteric Artery
Brief Title: Enucleation of Pancreatic Tumor by Blocking Abdominal Trunk and Superior Mesenteric Artery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Sheng Yan, Director, Head of Hepatology and Pancreatology, Principal Investigator, Clinical Professor., Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220492
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Tumor of Pancreas; Surgical Blood Loss
Keywords: Enucleation; pancreatic tumors; blood loss; the abdominal trunk; superior mesenteric artery
MeSH Terms: conditions — Pancreatic Neoplasms; Blood Loss, Surgical; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- blockade of arteries in laparoscopic pancreatic enucleation (Experimental): In the pancreatic enucleation, Kocher Maneuver was routinely performed at first. Then free the left side of the abdominal trunk and superior mesenteric artery, loose tissues easy to free.After Kocher Maneuver and other surgical procedures, the abdominal trunk and superior mesenteric artery exposed. Before resection of pancreatic tumors, a vascular occlusion clamp clip was used to block the root of both the abdominal trunk and superior mesenteric artery to control the pancreatic blood flow.
  Interventions: Procedure: blocking both the abdominal trunk and superior mesenteric artery in the pancreatic enucleation

INTERVENTIONS:
Procedure: blocking both the abdominal trunk and superior mesenteric artery in the pancreatic enucleation — In the pancreatic enucleation, Kocher Maneuver was routinely performed at first. Then free the left side of the abdominal trunk and superior mesenteric artery, loose tissues easy to free.After Kocher Maneuver and other surgical procedures, the abdominal trunk and superior mesenteric artery exposed. Before resection of pancreatic tumors, a vascular occlusion clamp clip was used to block the root of both the abdominal trunk and superior mesenteric artery to control the pancreatic blood flow.

SUMMARY:
Pancreatic enucleation could preserve more healthy pancreatic tissues and functions with a low recurrence risk. However, conventional enucleation can cause significant intraoperative bleeding, especially in which tumors in the pancreatic head, neck, and uncinate process of pancreas, as these tissues are rich in blood supply, mainly including the abdominal trunk and the superior mesenteric artery. In this study, we developed a novel method to control the pancreatic blood flow in laparoscopic enucleation--blocking the abdominal trunk and superior mesenteric artery with vascular occlusion clips in the process of resection, and evaluated its effectiveness and safety.

DETAILED DESCRIPTION:
Between March 2023 and May 2026, patients who underwent laparoscopic pancreatic enucleation by blocking both the abdominal trunk and superior mesenteric artery in the Second Affiliated Hospital of Zhejiang University would be included in our prospective study. Inclusion criteria: 1) benign or borderline tumors diagnosed pathologically, such as pancreatic neuroendocrine tumors, solid pseudopapillary tumors, and cystadenomas, without vascular invasion or distant metastasis;.2) tumors sited in the pancreatic head, neck, and uncinate process of pancreas; 3) blockade of both the abdominal trunk and superior mesenteric artery in the laparoscopic enucleation. Exclusion criteria:1) highly malignant pancreatic tumors, or tumors with infiltration or metastasis; 2) tumors of the body and tail of the pancreas;3) transfer to LPD or laparotomy. Patient characteristic including clinical, biochemical and radiological data will be recorded and analyzed. All patients will provide written informed consent before inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Benign or borderline tumors diagnosed pathologically, such as pancreatic neuroendocrine tumors, solid pseudopapillary tumors, and cystadenomas, without vascular invasion or distant metastasis
* Tumors sited in the pancreatic head, neck, and uncinate process of pancreas
* Blockade of both the abdominal trunk and superior mesenteric artery in the laparoscopic enucleation

Exclusion Criteria:

* Highly malignant pancreatic tumors, or tumors with infiltration or metastasis
* Tumors of the body and tail of the pancreas
* Transfer to LPD or laparotomy

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
blood loss | in the procedure
  blockade of both the abdominal trunk and superior mesenteric artery changes the blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhou, Dr., Principal Investigator — The Second Affiliated Hospital, Zhejiang Chinese Medical University
Locations (1):
- the Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD in the current study are available from central contact person upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will become available in June 2026 and for 6 months.
Access Criteria: The IPD in the current study are available from central contact person upon reasonable request.

REFERENCES:
- [Background] Song KB, Kim SC, Hwang DW, Lee JH, Lee DJ, Lee JW, Jun ES, Sin SH, Kim HE, Park KM, Lee YJ. Enucleation for benign or low-grade malignant lesions of the pancreas: Single-center experience with 65 consecutive patients. Surgery. 2015 Nov;158(5):1203-10. doi: 10.1016/j.surg.2014.10.008. Epub 2014 Nov 3. PMID 25633730
- See also: The aim of this study was to evaluate the postoperative clinical outcomes and long-term functional and oncologic results after pancreatic enucleation, and to compare the clinical results of laparoscopic and open enucleation. — https://pubmed.ncbi.nlm.nih.gov/25633730/